CLINICAL TRIAL: NCT05153512
Title: ADOlescent DysmenoRrhea Endometriosis Assessment Magnetic Resonance Imaging
Brief Title: ADOlescent DysmenoRrhea Endometriosis Assessment Magnetic Resonance Imaging (Adodream)
Acronym: Adodream
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A01354-51
Record Dates: First submitted 2021-11-25; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: MRI — Pelvic MRI without injection of contrast product and WITHOUT rectal or vaginal opacification

SUMMARY:
To date, no MRI study has been published describing the prevalence of endometriosis in adolescent girls, not even in those with significant dysmenorrhea and therefore more particularly at risk. Likewise, there are no precise data on the type of superficial or early-onset deep endometriosis that appears in adolescence. The collection of these data would allow an earlier diagnosis, because it is better documented, of endometriosis. The lesions would then be treated earlier, avoiding their development and the problems of infertility related to this pathology. The aim of this sudy is to assess the prevalence of endometriosis and its phenotypic representation in the study population consulting for dysmenorrhea with suspected endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 12 and 20 years old.
* After menarche.
* Requiring pelvic MRI for exploration of dysmenorrhea (after or not ultrasound), in the case of patients with suspected endometriosis, or for any other reason (cyst, tumor, non-obstructive urogenital malformations), in the case of patients without symptoms clinic associated with endometriosis.
* Patient affiliated or beneficiary of a social security scheme.
* Patient and her legal representative, if applicable, having been informed and not opposing this research.

Exclusion Criteria:

* Patient whose pelvic MRI is performed as part of an exploration of obstructive uterine malformations.
* Patient claustrophobic, making it impossible to perform an MRI.
* Contraindication to MRI: pacemaker, ferromagnetic object incompatible with MRI.
* Pregnant, breastfeeding or parturient woman.
* Protected patient: Major under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision; Hospitalized without consent.

Ages: 12 Years to 20 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Women between 12 and 20 years-old and suffering from dysmenorrhea
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2021-12-26 (Estimated)

PRIMARY OUTCOMES:
Number of patient with endometriosis detected on MRI | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- BLOMET clinic, Paris, IDF, France

REFERENCES:
- [Derived] Millischer AE, Santulli P, Da Costa S, Bordonne C, Cazaubon E, Marcellin L, Chapron C. Adolescent endometriosis: prevalence increases with age on magnetic resonance imaging scan. Fertil Steril. 2023 Apr;119(4):626-633. doi: 10.1016/j.fertnstert.2022.12.039. Epub 2022 Dec 31. PMID 36592649